CLINICAL TRIAL: NCT03670082
Title: Interventional, Open-label, Two-way Crossover, Single-dose Study Investigating the Absolute Bioavailability and Food Effect on the Pharmacokinetics of Lu AF35700 in Healthy Subjects
Brief Title: Study With Lu AF35700 in Healthy Men and Women in Fasting and Fed State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17482A
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — Lu AF35700

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Fasting condition in Period I (Experimental): Subjects will be in fasting condition in Period I and in a fed condition in Period II.
  Interventions: Drug: Lu AF35700; Drug: Lu AF35700 iv
- Group 2: Fed condition in Period I (Experimental): Subjects will be in fed condition in Period I and in fasting condition in Period II.
  Interventions: Drug: Lu AF35700

INTERVENTIONS:
Drug: Lu AF35700 — 20 mg Lu AF35700 single oral dose
Drug: Lu AF35700 iv — 100 μg [14C]-Lu AF35700 (4.7 μCi/174 kBq) single intravenous micro-dose
  Arms: Group 1: Fasting condition in Period I

SUMMARY:
The purpose of this study is to investigate the extent to which Lu AF35700 enters the bloodstream following pill intake and the influence of food on the uptake in healthy men and women

DETAILED DESCRIPTION:
Each subject will receive a single oral dose of Lu AF35700 on Day 1 in each Period. Subjects in Group 1 will be in fasting condition in Period I and in a fed condition in Period II. Subjects in Group 2 will be in fed condition in Period I and in fasting condition in Period II.

For Group 1, period 1 only, a single intravenous micro-dose of Lu AF35700 will be given 4 hours after oral dosing.

All subjects will be confined to the clinic from one day prior to the first dosing until Day 6 (120 hours post dose) for each dosing period. Periods I and II will be separated by a period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged ≥18 and ≤55 years
* Body Mass Index (BMI) of ≥18.5 and ≤30 kg/m2
* Subject must be in good general health as assessed using medical history, clinical laboratory tests, and physical examination

Exclusion Criteria:

* The subject must not be of childbearing potential (if a woman) or should use contraception, be surgically sterilized or not be sexually active (both sexes). Women must not be pregnant or lactating
* The subject must not be a CYP2D6 or a CYP2C19 poor metabolizer

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-01-13 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability Fabs | 0 to 120 hours
  Fabs= 100*(AUC0-72h, po*Div) / (AUC0-72h, iv*Dpo) (where D is the dose)

SECONDARY OUTCOMES:
AUC0-inf: area under the Lu AF35700 plasma concentration-time curve from zero to 72 hours | 0 to 120 hours
  Area under the plasma concentration-time curve from zero to 72 hours for Lu AF35700
Cmax: maximum observed plasma concentration | 0 to 120 hours
  Maximum observed plasma concentration of Lu AF35700
tmax: time at maximum observed plasma concentration | 0 to 120 hours
  Time at which maximum observed plasma concentration of Lu AF35700 occurred

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Covance, Leeds, United Kingdom